CLINICAL TRIAL: NCT04933487
Title: Prospective Evaluation of the Rotational Stability of the Ankoris Intraocular Lens
Brief Title: Rotational Stability Analysis of a Toric Monofocal IOL
Acronym: PHY2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY2013
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cataract; Lens Opacities; Astigmatism
Keywords: Intraocular Lens; Monofocal; Toric Lens
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankoris IOL Implantation experimental (Experimental): Monolateral implantation of toric intraocular lenses Ankoris
  Interventions: Device: IOL implantation experimental

INTERVENTIONS:
Device: IOL implantation experimental — Monolateral implantation of toric intraocular lenses Ankoris. (Manufactured by PhysIOL sa/nv, Liège, Belgium).

SUMMARY:
This is a single-center, prospective PMCF study whereby patients undergoing routine cataract surgery will have monolateral implantation of hydrophilic monofocal toric intraocular lens Ankoris.

DETAILED DESCRIPTION:
This is a single-center, prospective, nonrandomized PMCF study whereby patients undergoing routine cataract surgery will have monolateral implantation of hydrophilic monofocal toric intraocular lens (Ankoris). The device under investigation is manufactured by the sponsor of this study. The refractive power of the lens has a spherical and a cylindrical component. The IOLs will be implanted in the course of routine cataract surgery and will benefit to patients suffering from cataract development and showing pre-existing corneal astigmatism.

The primary objective of this study is to determine the rotational stability of the Ankoris intraocular lens. The secondary objective is to measure the residual astigmatism after Ankoris implantation with respect to the targeted astigmatism correction.

In total approx. 20 eyes of 20 patients will be recruited for this clinical study.

Follow-ups will be performed 1 day, 1 month, and 3 months after cataract surgery. Subjects would have the option for unscheduled visits if required medically.

ELIGIBILITY:
Inclusion Criteria:

* Cataracteous Eyes with no comorbidity
* Regular corneal astigmatism >1 dioptre and <3D determined by an automatic keratometer (regularity determined by the topography of the keratometry).
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent •>50 years old

Exclusion Criteria:

* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, Marfan's syndrome)
* Pupil abnormalitis (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Rotational stability - Photograph of IOL with dilated pupil to asses IOL rotation | 3 months postoperative
  Rotational stability of the ANKORIS is evaluated on the basis of slit-lamp photographies to capture the iris and the marks onto the lens. Descriptive statistics will be used to determine the IOL stability.

SECONDARY OUTCOMES:
Residual astigmatism after Ankoris implantation with respect to the targeted astigmatism correction. | Follow-ups will be performed 1 day, 1 month, and 3 months after cataract surgery
  Visual performance is determined in terms of monocular uncorrected distance visual acuity (UDVA), distance corrected visual acuity (DCVA) and postoperative refraction. Efficiency will be assessed using Alpins method.

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Dick, MD, Principal Investigator — Ruhr-Universitat Bochum, Bochum, Germany
Locations (1):
- Ruhr-Universitat Bochum, Bochum, Germany, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No